CLINICAL TRIAL: NCT02906592
Title: Using a Geriatric Oncology Assessment to Link With Services (GOAL)
Brief Title: Using a Geriatric Oncology Assessment to Link With Services
Acronym: GOAL
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Collaborators: Duke Cancer Institute (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00073547
Record Dates: First submitted 2016-09-15; First posted 2016-09-20 (Estimated); Last update posted 2018-01-11 (Actual); Status verified 2017-04

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No

SUMMARY:
The objective of this study is to implement a brief geriatric oncology assessment (GOA) in a community-based oncology clinic, the Scotland Cancer Treatment Center - a clinic within the Duke Cancer Network, located in the rural, low resource Scotland County community of North Carolina. Secondly, the investigators will evaluate the effectiveness of the brief GOA by comparing historical and post-GOA service referral patterns and adherence to planned cancer therapy. For this study, the investigators will prospectively enroll up to 60 patients who have been diagnosed and/or treated for cancer to complete the brief GOA. In addition to these 60 patients, the investigators will also conduct retrospective chart reviews on 120 patients that would be eligible for this study to evaluate past referral patterns. Eligible and consented patients will complete the brief GOA at the Scotland Cancer Treatment Center alongside their normal clinic appointment. The investigators will assess impact on the healthcare system by evaluating referral patterns (i.e., how many, what type of services) using the brief GOA data and EHR data. The study value includes the possibility for recognition and access to additional health care referrals if needed.

ELIGIBILITY:
Inclusion Criteria:

In order to be included in the project, patients must be:

1. Diagnosed for a solid tumor cancer (breast, lung, colon, rectal, colorectal (unspecified), pancreas, esophageal)
2. Diagnosis date within 12 months of identification
3. Receiving care at Scotland Cancer Treatment Center
4. Aged 60 years or older at the time of the visit
5. Planned therapy in the medical oncology clinic at the Scotland Cancer Treatment Center

Exclusion Criteria:

1. Diagnosis of metastatic cancer with <12 months life expectancy
2. Planned cancer therapy as surgery only
3. Receiving palliative or hospice care services (i.e., proxy for <12 months life expectancy)
4. Language (not proficient in English)
5. Nursing home/long-term care facility resident
6. Active diagnosis of psychosis (has been hospitalized in the last 30 days), schizophrenia, severe intellectual or developmental disabilities, or dementia
7. Patient deemed not fit/good candidate for study per provider recommendation

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Geriatric (60 years or older) patients in a community-based cancer clinic at Scotland Memorial Hospital. They serve a racially diverse (e.g., 35% African American, 10% Native American), elderly (e.g., 65% >65 years), rural, low resource community with over 20% of the population living in poverty.
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2017-01; Primary Completion 2017-09-29 (Actual); Study Completion 2017-09-29 (Actual)

PRIMARY OUTCOMES:
Change in referral patterns | retrospective data from 1/1/2013-7/7/2016
  Comparison of historical and post GOA service referral patterns
Time to complete the brief GOA | 6 months
Number of referrals completed | 6 months
Number of patients who needed help completing the brief GOA | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Leah Zullig, Ph.D., Principal Investigator — Duke University
Locations (1):
- Scotland Cancer Treatment Center, Laurinburg, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zullig LL, Kimmick G, Smith V, Little K, Bosworth HB, Gonzales S, Oakes MM, Shelby RA, Owen L, Altomare IP. Using a geriatric oncology assessment to link with services (GOAL). J Geriatr Oncol. 2019 Jan;10(1):164-168. doi: 10.1016/j.jgo.2018.06.004. Epub 2018 Jun 27. PMID 29958815